CLINICAL TRIAL: NCT06690268
Title: Multimodal Clinical-imaging-pathology-driven Artificial Intelligence Model for Predicting Postoperative Recurrence of Locally Advanced Gastric Cancer
Brief Title: Multimodal Model Predicts Recurrence
Acronym: FUTURE12
Status: Completed | Type: Observational
Sponsor: Qun Zhao (Other)
Responsible Party: Sponsor-Investigator, Qun Zhao, Professor, Hebei Medical University
Organization: Hebei Medical University (Other)
Other Study IDs: FUTURE12
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Gastric Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Multimodal AI-driven predictive model — This intervention involves a multimodal artificial intelligence (AI) model that integrates clinical data, imaging results, and pathology findings to predict the risk of postoperative recurrence in patients with locally advanced gastric cancer. Unlike traditional methods that may rely on single data sources, this AI-driven model synthesizes multiple types of patient information, offering a comprehensive and personalized prediction of recurrence risk. This approach aims to improve accuracy in identifying high-risk patients, allowing for more tailored follow-up and treatment planning to enhance patient outcomes.

SUMMARY:
This study focuses on developing an advanced model that combines clinical information, imaging, and pathology data to predict the likelihood of cancer returning after surgery in patients with locally advanced gastric cancer. By using artificial intelligence (AI), this model analyzes various data sources to create a more accurate prediction of recurrence risk, which can help doctors, patients, and families better understand the chances of recurrence. This AI-driven approach allows healthcare providers to make more informed decisions about personalized follow-up care and potential additional treatments to improve patient outcomes.

ELIGIBILITY:
**Inclusion Criteria:**

* Patients diagnosed with locally advanced gastric cancer (Stage II or III).
* Patients who have undergone surgical resection for gastric cancer.
* Patients with complete clinical, imaging, and pathology data available for analysis.
* Age 18 years or older.
* Patients who provide informed consent to participate in the study.

**Exclusion Criteria:**

* Patients with distant metastasis (Stage IV) at the time of diagnosis.
* Patients with incomplete or missing clinical, imaging, or pathology data.
* Patients who have received prior treatment for gastric cancer other than surgical resection.
* Patients with other concurrent malignancies.
* Patients who are unable or unwilling to comply with the study follow-up requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients (aged 18 and older) diagnosed with locally advanced gastric cancer (Stage II or III) who have undergone surgical resection. This population is selected based on the availability of complete clinical, imaging, and pathology data necessary for analysis by the multimodal AI-driven predictive model. The study focuses on assessing the postoperative recurrence risk in this specific group to improve personalized follow-up and treatment planning.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Prediction accuracy of postoperative recurrence in locally advanced gastric cancer | 24 months postoperative follow-up
  The primary outcome measure is the accuracy of the multimodal AI model in predicting the risk of postoperative recurrence in patients with locally advanced gastric cancer. This is assessed by comparing the model's predictions with actual recurrence events over a specified follow-up period, allowing evaluation of its effectiveness in identifying high-risk patients and guiding clinical decisions.

CONTACTS AND LOCATIONS:
Locations (1):
- the Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China